CLINICAL TRIAL: NCT02815982
Title: Targeting Caregivers to Enhance Health Behaviors in Pediatric Cancer Survivors (NOURISH-T)
Brief Title: Targeting Caregivers to Enhance Health Behaviors in Pediatric Cancer Survivors
Acronym: NOURISH-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: University of Pittsburgh (Other); Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R21CA167259-02 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2016-12

CONDITIONS: Obesity; Cancer
MeSH Terms: conditions — Obesity; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOURISH-T (Experimental): The intervention aims to increase caregivers' self-efficacy for behavioral change, and facilitate an authoritarian approach to parenting. Behavioral strategies such as self-monitoring, contingency management, and stimulus control are integrated in these sessions. Further, because participatory experiences enhance overall intervention efficacy, these activities are incorporated throughout, including self-assessments, discussions and experiential activities. Homework is assigned between sessions so skills can be practiced. We also focus on the caregivers' relationship with everyone in the family, not just the "identified patient" or overweight child.
  Interventions: Behavioral: NOURISH-T
- Enhanced Usual Care (Active Comparator): Caregivers randomized to the EUC will attend assessment sessions and an initial session moderated by an independent interventionist. The session addresses the role of diet and exercise in pediatric overweight. In addition, EUC caregivers receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Participants also receive a booster phone call 2 months after the end of the intervention period.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: NOURISH-T — Overweight/obesity family intervention
  Arms: NOURISH-T
Behavioral: Enhanced Usual Care — Publicly available overweight/obesity materials
  Arms: Enhanced Usual Care

SUMMARY:
This purpose of this pilot study is to investigate the feasibility of and optimal time post cancer treatment to offer caregivers a new health behavior change intervention (NOURISH-T), as well as assess its preliminary efficacy on specific child health behaviors. The study will also explore whether caregivers NOURISH-T exhibit more improvements than caregivers in EUC (standard care).

DETAILED DESCRIPTION:
Approximately 40% of off-treatment pediatric cancer survivors (PCS) are overweight or obese, which increases their risk for negative long-term physical health complications. Consistent with the Institute of Medicine's (IOM) emphasis on patients transitioning from treatment to cancer survivorship and increasing long-term healthy behaviors in these survivors, we conducted a pilot RCT to address the increasing overweight/obesity rates among PCS by targeting their caregivers as agents for PCS behavior change. We focused on parents' behaviors, attitudes and roles in promoting healthier eating and physical activity (PA) in PCS and adapted an evidence-informed, manualized parent intervention - NOURISH - found to be effective for parents of overweight and obese children and adolescents in reducing child and adolescent BMI. We adapted NOURISH for caregivers of 5 - 13 year old PCS (6 months -4 years off active cancer treatment). Our pilot feasibility RCT - NOURISH-T (Nourishing Our Understanding of Role modeling to Improve Support for Healthy Transitions) evaluates: 1) the preliminary feasibility efficacy of NOURISH-T for PCS, compared with an Enhanced Usual Care (EUC) control condition, and 2) factors to consider to improve future adaptations of the intervention. The project enrolled caregivers of PCS at two pediatric oncology clinics into the 6-week intervention (or EUC) with assessments of both caregivers and PCS occurring pre- and post-6 weeks of intervention, and at a 4-month follow-up. In comparison to EUC, we hypothesized that caregivers and PCS assigned to the NOURISH-T condition would show greater improvements in dietary intake, physical activity, and in anthropometric health indicators over time.

ELIGIBILITY:
Inclusion Criteria:

Caregivers

* Mothers and fathers (biologic/adoptive/step parents/legal guardians) of pediatric cancer survivors
* 18 years or older
* Fluent in English

Pediatric Cancer Survivors

* Diagnosis of cancer
* between 5-13 years of age at study entry
* off active cancer treatment for 6 months to 4 years,
* reside with a participating caregiver
* able to engage in PA tailored to current medical status
* NOT taking medications that affect body weight, e.g., steroids within 6 months of enrollment
* at or above the 85th BMI %ile.

Exclusion Criteria:

Caregivers

* are non-ambulatory
* do not reside with the PCS at least 50% of the time.

Pediatric cancer survivor

* relapse during the intervention
* taken a medication known to affect body weight such as oral steroids or antipsychotic medications within 6 months of enrollment

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Stern, PhD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stern M, Ewing L, Davila E, Thompson AL, Hale G, Mazzeo S. Design and rationale for NOURISH-T: a randomized control trial targeting parents of overweight children off cancer treatment. Contemp Clin Trials. 2015 Mar;41:227-37. doi: 10.1016/j.cct.2014.12.018. Epub 2015 Jan 2. PMID 25559916
- [Derived] Stern M, Bleck J, Ewing LJ, Davila E, Lynn C, Hale G, Mazzeo S. NOURISH-T: Targeting caregivers to improve health behaviors in pediatric cancer survivors with obesity. Pediatr Blood Cancer. 2018 May;65(5):e26941. doi: 10.1002/pbc.26941. Epub 2018 Jan 19. PMID 29350459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregivers and PCS were recruited as dyads, however, caregivers participated in the intervention (NOURISH-T vs EUC) and completed measures. PCS did not participate in the intervention and only completed measures. Outcomes are noted by whether caregivers or PCS completed measures.
Groups:
- NOURISH-T - Caregivers: Participants consisted of caregivers of obese pediatric cancer survivors (PCS). PCS are assessed at each time point (baseline, post intervention and 4 months follow-up), but do not directly participate in the intervention. NOURISH-T intervention aims to increase caregivers' self-efficacy for behavioral change, and facilitate an authoritarian approach to parenting. Behavioral strategies such as self-monitoring, contingency management, and stimulus control are integrated in these sessions. Further, because participatory experiences enhance overall intervention efficacy, these activities are incorporated throughout, including self-assessments, discussions and experiential activities. Homework is assigned between sessions so skills can be practiced. We also focus on the caregivers' relationship with everyone in the family, not just the "identified patient" or overweight child. Different measures are administered to caregivers and PCS.
  NOURISH-T: Overweight/obesity family intervention
- Enhanced Usual Care - Caregivers: Participants consisted of caregivers of obese pediatric cancer survivors (PCS). PCS are assessed but do not directly participate in the EUC group. randomized to the EUC attend assessment sessions and an initial session moderated by an independent interventionist. The session addresses the role of diet and exercise in pediatric overweight. In addition, EUC caregivers receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Participants also receive a booster phone call 2 months after the end of the intervention period. Different measures are administered to caregivers and PCS.
  Enhanced Usual Care: Publicly available overweight/obesity materials
- NOURISH-T - Pediatric Cancer Survivors (PCS): PCS are recruited with their caregivers, but do not participate in the intervention. PCS only complete measures.
- Enhanced Usual Care - Pediatric Cancer Survivors (PCS): PCS are recruited with their caregivers, but do not participate in the intervention (EUC), they only complete measures at each time point.
Period: Overall Study
Arm/Group | NOURISH-T - Caregivers | Enhanced Usual Care - Caregivers | NOURISH-T - Pediatric Cancer Survivors (PCS) | Enhanced Usual Care - Pediatric Cancer Survivors (PCS)
Started | 27 | 26 | 27 | 26
Completed (All participants completed at least baseline measurements) | 27 | 26 | 27 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We recruited caregivers as a function of their child's characteristics (e.g., PCS eligibility criteria of age, BMI percentile, time off active treatment)
Groups:
- NOURISH-T - Caregivers; NOURISH-T - Pediatric Cancer Survivors (PCS): The intervention aims to increase caregivers' self-efficacy for behavioral change, and facilitate an authoritarian approach to parenting. Behavioral strategies such as self-monitoring, contingency management, and stimulus control are integrated in these sessions. Further, because participatory experiences enhance overall intervention efficacy, these activities are incorporated throughout, including self-assessments, discussions and experiential activities. Homework will be assigned between sessions so skills can be practiced. We also focus on the caregivers' relationship with everyone in the family, not just the "identified patient" or overweight child.
  NOURISH-T: Overweight/obesity family intervention
- Enhanced Usual Care - Caregivers; Enhanced Usual Care - Pediatric Cancer Survivors (PCS): Caregivers randomized to the EUC will attend assessment sessions and an initial session moderated by an independent interventionist. The session will address the role of diet and exercise in pediatric overweight. In addition, EUC caregivers will receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Participants will also receive a booster phone call 2 months after the end of the intervention period.
  Enhanced Usual Care: Publicly available overweight/obesity materials
- Total: Total of all reporting groups
Arm/Group | NOURISH-T - Caregivers | NOURISH-T - Pediatric Cancer Survivors (PCS) | Enhanced Usual Care - Caregivers | Enhanced Usual Care - Pediatric Cancer Survivors (PCS) | Total
Number analyzed (Participants) | 27 | 27 | 26 | 26 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 27 | 0 | 26 | 53
  Between 18 and 65 years | 27 | 0 | 26 | 0 | 53
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  all Participants | 38.0 (8.4) | 9.48 (2.8) | 41.5 (9.2) | 10.48 (2.79) | 24.87 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 19 | 15 | 68
  Male | 6 | 14 | 7 | 11 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 4 | 16
  Not Hispanic or Latino | 20 | 20 | 17 | 17 | 74
  Unknown or Not Reported | 3 | 3 | 5 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1 | 2
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 20 | 20 | 17 | 17 | 74
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 8 | 8 | 28
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 26 | 26 | 106

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction and Exit Survey Composite Scale Score -- ONLY CAREGIVERS COMPLETED THIS MEASURE
Description: At the end of the final session (6-sessions), caregivers completed a likert-type survey assessing what they liked/disliked about the intervention, as well as what was/was not useful or helpful in reaching health goals. Eleven items were summed to obtain a total continuous composite satisfaction/liking score. Each item was measured on a likert scale ranging from strongly disagree (=1) to strongly agree (=5). The scale sum score ranged from 11 to 55 with higher scores indicating greater satisfaction with the intervention. More specifically, the higher the score, the more useful the caregiver thought the intervention and the more they liked participating in the intervention. Lower scores indicate that the caregiver thought the program was not useful and they did not like participating.
Time Frame: 6 weeks
Population: Independent Samples T-Test
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- NOURISH-T: The intervention aims to increase caregivers' self-efficacy for behavioral change, and facilitate an authoritarian approach to parenting. Behavioral strategies such as self-monitoring, contingency management, and stimulus control are integrated in these sessions. Further, because participatory experiences enhance overall intervention efficacy, these activities are incorporated throughout, including self-assessments, discussions and experiential activities. Homework is assigned between sessions so skills can be practiced. We also focus on the caregivers' relationship with everyone in the family, not just the "identified patient" or overweight child. PCS are assessed, but do not directly participate in the intervention.
  NOURISH-T: Overweight/obesity family intervention
- Enhanced Usual Care: Caregivers randomized to the enhanced usual care will attend assessment sessions and an initial session moderated by an independent interventionist. The session will address the role of diet and exercise in pediatric overweight. In addition, EUC caregivers will receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Caregivers also receive a booster phone call 2 months after the end of the intervention period. PCS are assessed, but do not directly participate in the intervention.
  Enhanced Usual Care: Publicly available overweight/obesity materials
Arm/Group | NOURISH-T | Enhanced Usual Care
Number analyzed (Participants) | 27 | 26
units on a scale | 46.2 (5.1) | 37.5 (8.1)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care; Test type: Superiority; p < .05, t-test, 2 sided; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-14.6 to -2.7]

2. Secondary Outcome: Automated Self-administered 24-Hour Dietary Recall (ASA 24) -- CAREGIVERS ONLY MEASURE
Description: A 24-hour recall was completed by caregivers using the Automated Self-administered 24-Hour Dietary Recall-2011 (adult version) at pre-intervention, post-intervention (6-weeks) and at 4 months follow-up. The outcome was measured as the number of calories consumed over 1-day. Caregivers reported detailed information on the foods consumed and quantity including the method used for preparation, portion sizes, and where the food was purchased using visual cues in the previous day through the ASA24 website (https://asa24.nci.nih.gov/). The website reported the total number of calories consumed based on the data input.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: calories
Groups:
- NOURISH-T: The intervention aims to increase caregivers' self-efficacy for behavioral change, and facilitate an authoritarian approach to parenting. Behavioral strategies such as self-monitoring, contingency management, and stimulus control are integrated in these sessions. Further, because participatory experiences enhance overall intervention efficacy, these activities are incorporated throughout, including self-assessments, discussions and experiential activities. Homework will be assigned between sessions so skills can be practiced. We also focus on the caregivers' relationship with everyone in the family, not just the "identified patient" or overweight child.
  NOURISH-T: Overweight/obesity family intervention
- Enhanced Usual Care (EUC): Caregivers randomized to the enhanced usual care will attend assessment sessions and an initial session moderated by an independent interventionist. The session will address the role of diet and exercise in pediatric overweight. In addition, EUC caregivers will receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Participants will also receive a booster phone call 2 months after the end of the intervention period.
  Enhanced Usual Care: Publicly available overweight/obesity materials
Arm/Group | NOURISH-T | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 27 | 26
calories
  Pre-Intervention | 1928.9 (628.9) | 1802.0 (641.3)
  Post-Intervention (6-weeks) | 1830.8 (818.7) | 1866.4 (732.6)
  Follow-up (4 Months) | 1732.6 (798.9) | 2012.2 (712.4)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care (EUC); We compared Post-intervention scores; Test type: Superiority; p < .001, t-test, 2 sided — p value was the actual signficance level; Mean Difference (Final Values) = 35.6, 95% CI 2-sided [-559.0 to 630.2]

3. Secondary Outcome: Child BMI Percentile -- ONLY Pediatric Cancer Survivors (PCS)
Description: Continuous child BMI percentile as a function of gender and age. This measure was obtained via the PCS medical chart.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: percentile
Groups:
- Enhanced Usual Care: Caregivers randomized to the enhanced usual care will attend assessment sessions and an initial session moderated by an independent interventionist. The session will address the role of diet and exercise in pediatric overweight. In addition, EUC caregivers will receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Participants will also receive a booster phone call 2 months after the end of the intervention period.
  Enhanced Usual Care: Publicly available overweight/obesity materials
Arm/Group | NOURISH-T | Enhanced Usual Care
Number analyzed (Participants) | 27 | 26
percentile
  Pre-Intervention | 95.3 (3.9) | 95.9 (4.1)
  Post-Intervention (6-weeks) | 95.2 (3.9) | 95.7 (4.7)
  Follow-up (4 Months) | 94.8 (3.2) | 93.4 (5.1)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care; We compared Post-intervention BMI; Test type: Superiority; p < .001, t-test, 2 sided — controlling for caregiver BMI at baseline and PCS BMI percentile at baseline; Mean Difference (Final Values) = .47, 95% CI 2-sided [-2.3 to 3.3]

4. Secondary Outcome: Child Sugar Sweet Beverage and Fast Food Intake Scale Sum Score -- ONLY Pediatric Cancer Survivors (PCS) Assessed on This Measure
Description: This 8-item questionnaire was completed by the pediatric cancer survivor and assessed child intake of sugar sweetened beverages, breakfast and dinner habits, as well as frequency of fast food intake. The sum score represents the total number of sugary beverages consumed and the number of times consuming fast food in the prior week. Higher scores indicate greater consumption of sugary beverages and fast food in the prior week. The sum score could range from 0 and has no upper limit.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enhanced Usual Care(EUC): Caregivers randomized to the enhanced usual care will attend assessment sessions and an initial session moderated by an independent interventionist. The session will address the role of diet and exercise in pediatric overweight. In addition, EUC caregivers will receive nationally available print or web-based brochures on pediatric overweight on 2 occasions during the study so that similar (but not as intensive) information is provided in the intervention and EUC arms of the study. Participants will also receive a booster phone call 2 months after the end of the intervention period.
  Enhanced Usual Care: Publicly available overweight/obesity materials
Arm/Group | NOURISH-T | Enhanced Usual Care(EUC)
Number analyzed (Participants) | 27 | 26
units on a scale
  Pre-Intervention | 9.4 (7.3) | 9.5 (7.4)
  Post-Intervention (6-weeks) | 7.8 (5.0) | 7.7 (7.5)
  Follow-up (4 Months) | 5.1 (4.4) | 7.3 (3.3)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care(EUC); We compared Post-intervention scores; Test type: Superiority; p < .03, t-test, 2 sided — p < .05 was the threshold; Mean Difference (Final Values) = -.12, 95% CI 2-sided [-5.4 to 5.2]

5. Secondary Outcome: Child Feeding Questionnaire Sum Score -- ONLY CAREGIVERS COMPLETED THIS MEASURE
Description: This 31-item questionnaire assesses parental approaches to and attitudes about feeding their children. Sub-scales include concerns about child weight, monitoring, restriction, and pressure to eat. The sum score of the Likert items ranged from 31 to 155 with higher scores indicating greater perceived concern, monitoring, restriction and pressure to eat.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOURISH-T | Enhanced Usual Care(EUC)
Number analyzed (Participants) | 27 | 26
units on a scale
  Pre-Intervention | 97.3 (15.2) | 96.7 (13.6)
  Post-Intervention (6-weeks) | 95 (10.9) | 98.5 (10.2)
  Follow-up (4 Months) | 95.2 (11.5) | 92.3 (7.9)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care(EUC); Test type: Superiority; p < .09, t-test, 2 sided — p < .05 was threshold; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-4.3 to 11.3]

6. Secondary Outcome: Number of Daily Steps Averaged Over a Week -- ONLY Pediatric Cancer Survivors (PCS) Assessed
Description: PCS and caregivers were trained to wear a piezoelectric, computer downloadable pedometer consecutively for 7 days prior to the pre- and post- intervention and 4 months post-intervention assessments to assess frequency of daily steps. The scale was measured as the continuous number of daily steps averaged over a week.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: Average number of steps per day
Arm/Group | NOURISH-T | Enhanced Usual Care(EUC)
Number analyzed (Participants) | 27 | 26
Average number of steps per day
  Pre-Intervention | 5695.5 (2448.5) | 6568.4 (2238.9)
  Post-Intervention (6-weeks) | 6279.4 (3582.9) | 5950.8 (2502.2)
  Follow-up (4 Months) | 7162.6 (2123.7) | 8674.7 (3143.9)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care(EUC); We compared Post-intervention scores; Test type: Superiority; p < .08, t-test, 2 sided — p < .05 threshold,; Mean Difference (Final Values) = -328.6, 95% CI 2-sided [-2868.4 to 2211.2]

7. Secondary Outcome: Child Waist to Hip Ratio -- ONLY Pediatric Cancer Survivors (PCS) ASSESSED
Description: Measured at the clinic via standardized equipment.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | NOURISH-T | Enhanced Usual Care
Number analyzed (Participants) | 27 | 26
ratio
  Pre-Intervention | .94 (.1) | .97 (.1)
  Post-Intervention (6-weeks) | .93 (.05) | .98 (.08)
  Follow-up (4 Months) | .92 (.09) | .99 (.08)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care; We compared Post-intervention scores; Test type: Superiority; p < .0001, t-test, 2 sided — threshold set at p < .05; Mean Difference (Final Values) = .06, 95% CI 2-sided [.01 to .11]

8. Secondary Outcome: Parent BMI Score -- CAREGIVER MEASURE
Description: Measured at the clinic via standardized equipment.
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | NOURISH-T | Enhanced Usual Care
Number analyzed (Participants) | 27 | 26
kg/m^2
  Pre-Intervention | 32.9 (12.2) | 32.1 (6.4)
  Post-Intervention (6-weeks) | 33.2 (13.5) | 30.3 (6.6)
  Follow-up (4 Months) | 32.4 (9.5) | 32.5 (8.2)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care; We compared Post-intervention scores; Test type: Superiority; p < .001, t-test, 2 sided — threshold set at p < .05; Mean Difference (Final Values) = -2.85, 95% CI 2-sided [-11.3 to 5.65]

9. Secondary Outcome: Parent Waist to Hip Ratio -- CAREGIVER MEASURE
Description: Measured at the clinic via standardized equipment
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | NOURISH-T | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 27 | 26
ratio
  Pre-Intervention | .94 (.06) | .91 (.09)
  Post-Intervention (6-weeks) | .90 (.06) | .91 (.06)
  Follow-up (4 Months) | .90 (.05) | .94 (.07)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care (EUC); We compared Post-intervention scores; Test type: Superiority; p < .001, t-test, 2 sided — threshold p < .05; Mean Difference (Final Values) = .01, 95% CI 2-sided [-.04 to .06]

10. Secondary Outcome: Number of Daily Steps Averaged Over a Week for Caregivers -- CAREGIVER MEASURE
Description: as for outcome 6
Time Frame: Pre-Intervention, Post-Intervention (6-weeks), Follow-up (4 Months)
Measure: Mean (Standard Deviation); unit: Average number of steps per day
Arm/Group | NOURISH-T | Enhanced Usual Care
Number analyzed (Participants) | 27 | 26
Average number of steps per day
  Pre-Interve'ntion | 7016.7 (2928.3) | 6288.3 (2923.2)
  Post-Intervention (6-weeks) | 5439.0 (3441.7) | 5090.1 (1893.8)
  Follow-up (4 Months) | 7087.4 (4506.1) | 5891.2 (2205.2)
Statistical Analysis 1: Comparison: NOURISH-T vs Enhanced Usual Care; We compared Post-intervention scores; Test type: Superiority; p < .12, t-test, 2 sided — p < .05 was the threshold; Mean Difference (Final Values) = -348.9, 95% CI 2-sided [-2762.5 to 2064.8]

ADVERSE EVENTS:
Time Frame: 2 years monitored for both the caregivers and for the pediatric cancer survivors (PCS); none identified
Arm/Group | NOURISH-T - Caregivers | Enhanced Usual Care - Caregivers | NOURISH-T - Pediatric Cancer Survivors (PCS) | Enhanced Usual Care - Pediatric Cancer Survivors (PCS)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/27 | 0/26

LIMITATIONS AND CAVEATS:
Self-report nature of the measures; Measurement error associated with the use of the pedometers; Differences in protocol between sites impacted sample size. Dyads were recruited, different measures were administered to caregivers and PCS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes